CLINICAL TRIAL: NCT07129824
Title: Relationship Between Eating Habits, Food Preferences and Symptoms in Chronic Gastritis Patients
Brief Title: Relationship Between Diet and Gastritis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ola Abdelmohsen Fathy, Family medicine resident at Sohag Health Directorate, Sohag University
Other Study IDs: Soh-Med--25-7-2MS
Record Dates: First submitted 2025-08-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Gastritis
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic gastritis patients: Adults aged 18 years or above with gastrointestinal symptoms for a week or longer exclude who reported having other digestive system diseases such as peptic ulcer, pancreatitis, hepatitis, and cirrhosis also serious heart, brain, liver, kidney and hematopoietic system dysfunction. Severe mental illness (such as schizophrenia, depression, and anxiety), and food or drug allergies, pregnancy, or breastfeeding and symptoms that occurred after taking prescription or over-the-counter drugs, especially aspirin or other pain relievers are also excluded
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe the effect of eating habits and food preferences on symptoms of chronic gastritis

SUMMARY:
Chronic gastritis (CG) is a prevalent and persistent inflammatory condition that affects the gastric mucosa, carrying a significant global burden. Although CG may remain asymptomatic in some cases, many patients experience gastrointestinal (GI) symptoms such as epigastric pain, bloating, nausea, vomiting, and appetite loss.

Diet plays a crucial role in both the development and progression of CG. there is a significant relationship between dietary behaviors, GI symptoms, and quality of life (QoL) in CG patients. Poor dietary habits have been associated with increased symptom severity, while healthier eating behaviors correlate with better physical and mental well-being.

Most research has focused on dietary risk factors in gastric cancer patients, with limited studies exploring their impact on CG and its symptoms. Furthermore, while nutritional adjustments are frequently recommended in clinical practices such as reducing coffee and alcohol intake and avoiding heavy smoking, there is a lack of comprehensive studies evaluating the relationship between eating habits, food preferences, and symptom severity in CG patients

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18 years or above

  * All consecutive patients with gastrointestinal symptoms for a week or longer.

Exclusion Criteria:

* Subjects who reported having other digestive system diseases such as peptic ulcer, pancreatitis, hepatitis, and cirrhosis
* Serious heart, brain, liver, kidney, or hematopoietic system dysfunction or other serious diseases
* Severe mental illness (such as schizophrenia, depression, and anxiety)
* Food or drug allergies, pregnancy, or breastfeeding
* Symptoms that occurred after taking prescription or over-the-counter drugs, especially aspirin or other pain relievers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or above with gastrointestinal symptoms for a week or longer.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
measure the percentage of patients with chronic gastritis who follow unhealthy dietary habits. | 12 months
  measure the percentage of patients with chronic gastritis who follow unhealthy dietary habits by standardized questionnaire consisted of three main sections:
  1. Sociodemographic Characteristics (age, sex, educational level, height, and weight).
  2. Gastrointestinal Symptoms (stomachache, gastric distention, hiccup, belching, heartburn, acid reflux, abdominal bloating, nausea, abdominal pain, vomiting, diarrhea, early satiety, appetite changes, food intake quantity, and symptom-related triggers)
  3. Dietary Factors (eating habits, food preferences)

CONTACTS AND LOCATIONS:
Overall Officials: Ola A fathy, Family medicine resident, Principal Investigator — Sohag University
Locations (1):
- Sohag university hospitals, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azer SA, Awosika AO, Akhondi H. Gastritis. 2024 Jun 22. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK544250/ PMID 31334970